CLINICAL TRIAL: NCT04918927
Title: Favipiravir and/or Nitazoxanide: a Randomized, Double-blind, Placebo-controlled Trial of Early Antiviral Therapy in COVID-19 (FANTAZE)
Brief Title: Favipiravir +/- Nitazoxanide: Early Antivirals Combination Therapy in COVID-19
Acronym: FANTAZE
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Coordinación de Investigación en Salud, Mexico (Other Government)
Collaborators: University College, London (Other); Centro de Investigacion y Estudios Avanzados del Instituto Politecnico Nacional (CINVESTAV) (Unknown); Universidad Autonoma de Guadalajara (Unknown); Siegfried Rhein S.A. de C.V. (Unknown); Strides Pharma Science Limited (Unknown); Hakken Enterprise (Unknown)
Responsible Party: Principal Investigator, Jorge Escobedo de la Pena, Head of the Epidemiology Clinical Research Unit, Coordinación de Investigación en Salud, Mexico
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2021-785-018
Record Dates: First submitted 2021-06-04; First posted 2021-06-09 (Actual); Last update posted 2023-03-24 (Actual); Status verified 2023-03

CONDITIONS: Covid19
MeSH Terms: conditions — COVID-19 | interventions — favipiravir; nitazoxanide

STUDY DESIGN:
Intervention Model Description: Phase IIA randomised, double-blind, placebo-controlled, interventional trial.
Who Masked: Participant, Care Provider, Investigator
Masking Description: Double-blind
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arm 1: Favipiravir + Nitazoxanide (Experimental): Oral Favipiravir 1800 mg twice daily on Day 1, followed by 400 mg four (4) times daily from Day 2 to Day 7 PLUS Nitazoxanide at 1000 mg twice daily on Day 1 followed by 500 mg four (4) times daily from Day 2 to Day 7
  Interventions: Drug: Favipiravir; Drug: Nitazoxanide
- Arm 2: Favipiravir + Nitazoxanide placebo (Experimental): Oral favipiravir, 1800 mg twice daily on Day 1, followed by 400 mg four (4) times daily from Day 2 to Day 7 PLUS Nitazoxanide matched placebo at 1000 mg twice daily on Day 1 followed by 500 mg four (4) times daily from Day 2 to Day 7.
  Interventions: Drug: Favipiravir; Other: Nitazoxanide Placebo

INTERVENTIONS:
Drug: Favipiravir — Oral Favipiravir 1800 mg twice daily on Day 1, followed by 400 mg four (4) times daily from Day 2 to Day 7
Drug: Nitazoxanide — Nitazoxanide at 1000 mg twice daily on Day 1 followed by 500 mg four (4) times daily from Day 2 to Day 7
  Other Names: Daxon
  Arms: Arm 1: Favipiravir + Nitazoxanide
Other: Nitazoxanide Placebo — Nitazoxanide matched placebo at 1000 mg twice daily on Day 1 followed by 500 mg four (4) times daily from Day 2 to Day 7.
  Other Names: Daxon Placebo
  Arms: Arm 2: Favipiravir + Nitazoxanide placebo

SUMMARY:
The 2020 pandemic of SARS-CoV-2 causing COVID-19 disease is an unprecedented global emergency. COVID-19 appears to be a disease with an early phase where the virus replicates, coinciding with first presentation of symptoms, followed by a later 'inflammatory' phase which results in severe disease in some individuals. It is known from other rapidly progressive infections such as sepsis and influenza that early treatment with antimicrobials is associated with better outcome. The hypothesis is that this holds for COVID-19 and that early antiviral treatment may prevent progression to the later phase of the disease.

The plan is to conduct a proof-of-principle placebo-controlled clinical trial of favipiravir plus or minus nitazoxanide in health workers, their household members and IMSS beneficiaries. Participants with or without symptomatic COVID-19 or tested positive will be assigned to receive favipiravir plus nitazoxanide or favipiravir plus nitazoxanide placebo. The primary outcome will be the difference in the amount of virus ('viral load') in the upper respiratory tract after 5 days of therapy. Secondary outcomes will include hospitalization, major morbidity and mortality, pharmacokinetics, and impact of antiviral therapy on viral genetic mutation rate.

If favipiravir with nitazoxanide demonstrates important antiviral effects without significant toxicity, there will be a strong case for a larger trial in people at high risk of hospitalization or intensive care admission, for example older patients and/or those with comorbidities and with early disease.

DETAILED DESCRIPTION:
FANTAZE is a Phase IIA randomised, double-blind, placebo-controlled, interventional trial.Participants will be adults who have developed the early symptoms of COVID-19 within the first 5 days, or tested positive for SARS-CoV-2 within the first 7 days of symptom onset, or not presenting symptoms but tested positive within the last 48 hours (date/time of test must be within 48 hours of enrolment).

Eligible participants will be randomised 1:1 to receive one of the following combinations:

Favipiravir + Nitazoxanide (both active); Favipiravir active + Nitazoxanide placebo;

All participants will be enrolled and followed up for 28 days. A saliva sample for virological analysis and safety blood samples will be collected at baseline, as well as a diagnostic nose and throat swab, if the participant hasn't been tested for COVID-19 yet. Following randomisation, participants will take trial medication for 7 days and during this period will take a daily saliva sample and complete a symptoms diary including four daily temperature measurements.

Participants will have two follow-up visits at Day 7 and Day 14 where they will be assessed and undergo blood tests for toxicity and pharmacokinetic assessment (on Day 7 only) and provide stool samples. Participants will have a telephone follow up three (3) weeks after their last day of treatment (Day 7) and further information will be collected through a questionnaire.

ELIGIBILITY:
Inclusion Criteria:

1. Health workers, their household members and, IMSS beneficiaries with the following:

   * Symptoms compatible with COVID-19 disease (Fever >37.8oC on at least one occasion AND either cough and/ or anosmia) within the first 5 days of symptom onset (date/time of enrolment must be within the first 5 days of symptom onset)
   * OR ANY symptoms compatible with COVID-19 disease (may include, but are not limited to fever, cough, shortness of breath, malaise, myalgia, headache, coryza) and tested positive for SARS-CoV-2 within the first 7 days of symptom onset (date/time of enrolment must be within the first 7 days of symptom onset)
   * OR no symptoms but tested positive for SARS-CoV-2 within the last 48 hours (date/time of test must be within 48 hours of enrolment)
2. Male or female aged 18 years to 70 years old inclusive at screening
3. Willing and able to take daily saliva samples
4. Able to provide full informed consent and willing to comply with trial-related procedures

Exclusion Criteria:

1. Known hypersensitivity to any of the active ingredients or excipients in favipiravir, and in nitazoxanide and matched placebo
2. Chronic liver disease at screening (known cirrhosis of any aetiology, chronic hepatitis (e.g. autoimmune, viral, steatohepatitis), cholangitis or any known elevation of liver aminotransferases with AST or ALT > 3 X ULN)*
3. Chronic kidney disease (stage 3 or beyond) at screening: eGFR < 60 ml/min/1.73m2*
4. HIV infection, if untreated, detectable viral load or on protease inhibitor therapy
5. Any clinical condition which the investigator considers would make the participant unsuitable for the trial
6. Concomitant medications known to interact with favipiravir, and with nitazoxanide and matched placebo, and carry risk of toxicity for the participant (See Appendix 4)
7. Current severe illness requiring hospitalisation
8. Pregnancy and/ or breastfeeding
9. Eligible female participants of childbearing potential and male participants with a partner of childbearing potential not willing to use highly effective contraceptive measures during the trial and within the time point specified following last trial treatment dose.
10. Participants enrolled in any other interventional drug or vaccine trial (co-enrolment in observational studies is acceptable).

    * Considering the importance of early treatment of COVID-19 to impact viral load, the absence of chronic liver/ kidney disease will be confirmed verbally by the participant during pre- screening and Screening/Baseline visit. Safety blood samples will be collected at Screening/Baseline visit (Day 1) and test results will be examined as soon as they become available within 24 hours.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2021-10-12 (Actual); Primary Completion 2023-03-21 (Actual); Study Completion 2023-03-21 (Actual)

PRIMARY OUTCOMES:
Upper respiratory tract viral load at Day 5. | Day 5 from randomisation
  Quantitative polymerase chain reaction (PCR) performed on saliva samples at Day 5 of therapy

SECONDARY OUTCOMES:
Percentage of participants with undetectable upper respiratory tract viral load after 5 days of therapy | Day 5 from randomisation
  Method of measurement: quantitative polymerase chain reaction (PCR) performed on saliva samples.
Proportion of participants with undetectable stool viral load after 7 days of therapy and 14 days post-randomisation. | Day 7 and Day 14 from randomization
  Method of measurement: PCR performed on stool samples
Rate of decrease in upper respiratory tract viral load during 7 days of therapy. | From day of randomisation to day 7
  Method of measurement: PCR performed on daily saliva samples
Duration of fever following commencement of medication | From day of randomisation to day 7
  Methods of measurement: daily body temperature records between Day 1 and Day 7 post-randomisation
Proportion of participants with hepatotoxicity after 7day of therapy and 14 days post-randomisation. | Day 7 and day 14 from randomisation.
  Method of measurement: standard diagnostic laboratory assays for liver transaminases, alkaline phosphatase and bilirubin.
Proportion of participants with other medication-related toxicity after 7 days of therapy and 14 days post-randomisation. | Day 7 and Day 14 from randomisation.
  Methods of measurement: determination of medication-related adverse events by investigators.
Proportion of participants admitted to hospital with COVID-19 related illness. | 28 days from randomisation.
  Methods of measurement: participant self-report, review of hospital records and discharge summaries
Proportion of participants admitted to ICU with COVID-19 related illness. | 28 days from randomisation.
  Methods of measurement: participant self-report, review of hospital records and discharge summaries.
Proportion of participants who have died with COVID-19 related illness | 28 days from randomisation.
  Methods of measurement: next of kin report, review of hospital records and discharge summaries.
Pharmacokinetic analysis of favipiravir and tizoxanide: Clearance (CL) | Day 7 from randomization
  Methods of measurement: assay of favipiravir and tizoxanide levels in plasma at Day 7 of therapy. All participants from each arm will provide a pre-dose sample and two post-dose (30 to 60 min) samples on Day 7 of therapy. A nonlinear mixed effects model will be fitted jointly to favipiravir and tizoxanide pharmacokinetic data.
  The model will estimate the following primary PK parameter: Clearance (CL).
Pharmacokinetic analysis of favipiravir and tizoxanide: Volume of distribution (V) | Day 7 from randomization
  Methods of measurement: assay of favipiravir and tizoxanide levels in plasma at Day 7 of therapy. All participants from each arm will provide a pre-dose sample and two post-dose (30 to 60 min) samples on Day 7 of therapy. A nonlinear mixed effects model will be fitted jointly to favipiravir and tizoxanide pharmacokinetic data.
  The model will estimate the following primary PK parameter: Volume of distribution (V),
Pharmacokinetic analysis of favipiravir and tizoxanide: Absorption rate constant (Ka) | Day 7 from randomization
  Methods of measurement: assay of favipiravir and tizoxanide levels in plasma at Day 7 of therapy. All participants from each arm will provide a pre-dose sample and two post-dose (30 to 60 min) samples on Day 7 of therapy. A nonlinear mixed effects model will be fitted jointly to favipiravir and tizoxanide pharmacokinetic data.
  The model will estimate the following primary PK parameter: Absorption rate constant (Ka).
Pharmacokinetic analysis of favipiravir and tizoxanide: Maximum concentration (Cmax) | Day 7 from randomization
  Methods of measurement: assay of favipiravir and tizoxanide levels in plasma at Day 7 of therapy. All participants from each arm will provide a pre-dose sample and two post-dose (30 to 60 min) samples on Day 7 of therapy. A nonlinear mixed effects model will be fitted jointly to favipiravir and tizoxanide pharmacokinetic data.
  The model will estimate the previous described primary PK parameters from which the following secondary parameter will be derived: Maximum concentration (Cmax),
Pharmacokinetic analysis of favipiravir and tizoxanide: Time to maximum concentration (Tmax) | Day 7 from randomization
  Methods of measurement: assay of favipiravir and tizoxanide levels in plasma at Day 7 of therapy. All participants from each arm will provide a pre-dose sample and two post-dose (30 to 60 min) samples on Day 7 of therapy. A nonlinear mixed effects model will be fitted jointly to favipiravir and tizoxanide pharmacokinetic data.
  The model will estimate the previous described primary PK parameters from which the following secondary parameter will be derived: Time to maximum concentration (Tmax),
Pharmacokinetic analysis of favipiravir and tizoxanide: Elimination rate constant (Ke) | Day 7 from randomization
  Methods of measurement: assay of favipiravir and tizoxanide levels in plasma at Day 7 of therapy. All participants from each arm will provide a pre-dose sample and two post-dose (30 to 60 min) samples on Day 7 of therapy. A nonlinear mixed effects model will be fitted jointly to favipiravir and tizoxanide pharmacokinetic data.
  The model will estimate the previous described primary PK parameters from which the following secondary parameter will be derived: Elimination rate constant (Ke),
Pharmacokinetic analysis of favipiravir and tizoxanide: Area Under the Curve extrapolated to infinity (AUC 80-inf). | Day 7 from randomization
  Methods of measurement: assay of favipiravir and tizoxanide levels in plasma at Day 7 of therapy. All participants from each arm will provide a pre-dose sample and two post-dose (30 to 60 min) samples on Day 7 of therapy. A nonlinear mixed effects model will be fitted jointly to favipiravir and tizoxanide pharmacokinetic data.
  The model will estimate the previous described primary PK parameters from which the following secondary parameter will be derived:
  Area Under the Curve extrapolated to infinity (AUC 80-inf)),
Pharmacodynamic analysis of favipiravir and tizoxanide: Rate of viral load decline (delta) | Day 7 from randomization
  A nonlinear mixed effects model will be fitted jointly to favipiravir and tizoxanide pharmacokinetic and viral load (pharmacodynamic) data.
  The model will estimate the following pharmacodynamic parameter: Rate of viral decline (delta) Maximum increase in viral load under drug treatment (Emax), Concentration to achieve half the maximum possible effects (EC50)
Pharmacodynamic analysis of favipiravir and tizoxanide: Maximum increase in viral load under drug treatment (Emax). | Day 7 from randomization
  A nonlinear mixed effects model will be fitted jointly to favipiravir and tizoxanide pharmacokinetic and viral load (pharmacodynamic) data.
  The model will estimate the following pharmacodynamic parameter: Maximum increase in viral load under drug treatment (Emax).
Pharmacodynamic analysis of favipiravir and tizoxanide: Concentration to achieve half the maximum possible effects (EC50) | Day 7 from randomization
  A nonlinear mixed effects model will be fitted jointly to favipiravir and tizoxanide pharmacokinetic and viral load (pharmacodynamic) data.
  The model will estimate the following pharmacodynamic parameter: Concentration to achieve half the maximum possible effects (EC50)
Exploratory: proportion of participants with deleterious or resistance-conferring mutations in SARS-CoV-2. | Day 7 from randomization
  Method of measurement: deep sequencing of virus and bioinformatic analysis.

CONTACTS AND LOCATIONS:
Overall Officials: Jorge Escobedo, Dr., Principal Investigator — Instituto Mexicano del Seguro Social
Locations (1):
- Hospital de Infectología "Daniel Méndez Hernández" del Centro Médico Nacional La Raza, Mexico City, Azcapotzalco, Mexico

IPD SHARING:
Plan to Share IPD: Undecided
No plan to share IPD has been made at this time

REFERENCES:
- [Derived] Smith T, Hoyo-Vadillo C, Adom AA, Favari-Perozzi L, Gastine S, Dehbi HM, Villegas-Lara B, Mateos E, Gonzalez YSP, Navarro-Gualito MD, Cruz-Carbajal AS, Cortes-Vazquez MA, Bekker-Mendez C, Aguirre-Alvarado C, Aguirre-Gil G, Delgado-Pastelin L, Owen A, Lowe D, Standing J, Escobedo J. Favipiravir and/or nitazoxanide: a randomized, double-blind, 2x2 design, placebo-controlled trial of early therapy in COVID-19 in health workers, their household members, and patients treated at IMSS (FANTAZE). Trials. 2022 Jul 22;23(1):583. doi: 10.1186/s13063-022-06533-0. PMID 35869526